CLINICAL TRIAL: NCT02538445
Title: Can we Forget? Directed Forgetting and Embodied Cognition in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1001156; 2010-A01372-37 (Other: ANSM)
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2015-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Memory; Cognition
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Patients group 1 (Experimental): Memorization of the verbs by miming the action
  Interventions: Other: Memorization of the verbs by miming the action
- Patients group 2 (Experimental): Memorization of the verbs by imagining the action
  Interventions: Other: Memorization of the verbs by imagining the action
- Patients group 3 (Experimental): Memorization of the action verbs by means of another word
  Interventions: Other: Memorization of the action verbs by means of another word
- Patients group 4 (Experimental): Simple memorization of the verbs
  Interventions: Other: Simple memorization of the verbs
- Healthy volonteers group 1 (Active Comparator): Memorization of the verbs by miming the action
  Interventions: Other: Memorization of the verbs by miming the action
- Healthy volonteers group 2 (Active Comparator): Memorization of the verbs by imagining the action
  Interventions: Other: Memorization of the verbs by imagining the action
- Healthy volonteers group 3 (Active Comparator): Memorization of the action verbs by means of another word
  Interventions: Other: Memorization of the action verbs by means of another word
- Healthy volonteers group 4 (Active Comparator): Simple memorization of the verbs
  Interventions: Other: Simple memorization of the verbs

INTERVENTIONS:
Other: Memorization of the verbs by miming the action — The participant reads aloud the verbs that appear on the screen, by performing the corresponding action verb.
  Arms: Healthy volonteers group 1; Patients group 1
Other: Memorization of the verbs by imagining the action — The participant reads aloud the verbs that appear on the screen, by imagining the corresponding action verb.
  Arms: Healthy volonteers group 2; Patients group 2
Other: Memorization of the action verbs by means of another word — The participant reads aloud the verbs that appear on the screen. Then, he reads, without memorizing it, a word associated with the action verb to be learnt to favor the memorization of that one. The word is written near the action verb.
  Arms: Healthy volonteers group 3; Patients group 3
Other: Simple memorization of the verbs — The participant reads aloud the verbs that appear on the screen, without additional instructions (control condition).
  Arms: Healthy volonteers group 4; Patients group 4

SUMMARY:
Based on the theory of embodied cognition, which focuses on the influence of sensory and motor processes on cognition, researchers propose to study the influence of the action on memorization and inhibition in patients suffering from schizophrenia, using a directed forgetting paradigm. The directed forgetting paradigm is used, composed of two lists of action verbs. The instruction "to forget" is given at the end of learning the first list (To Be Forgotten (TBF)), following a simulation of a computer bug. Therefore a second list is presented to be learned and remembered (To Be Remembered (TBR)). A recognition task is performed at the end. The action verbs had to be encoded using four conditions: action performed, mimed, imagined action, action with a contextual word, reading the action verb only. 48 schizophrenic patients were included in this study. Patients were randomized to have 10 participants per condition. 48 controls matched by age, gender, laterality and education are also included and randomized in the same modality. This study aims to show that the encoding of sensory-motor components, more than providing a context could improve the inhibitory capacities but also memory in schizophrenia, and possibly be used in remediation cognitive.

DETAILED DESCRIPTION:
Researchers used the directed forgetting paradigm composed of two lists of action verbs. The instruction "to forget" is given at the end of learning the first list (To Be Forgotten (TBF)), following a simulation of a computer bug. Therefore a second list is presented to be learned and remembered (To Be Remembered (TBR)). A recognition task is performed at the end. The action verbs had to be encoded using four conditions: action performed, mimed, imagined action, action with a contextual word, reading the action verb only. 48 schizophrenic patients were included in this study. Patients were randomized to have 10 participants per condition. 48 controls matched by age, gender, laterality and education are also included and randomized in the same modality. This study aims to show that the encoding of sensory-motor components, more than providing a context could improve the inhibitory capacities but also memory in schizophrenia, and possibly be used in remediation cognitive.

ELIGIBILITY:
Inclusion Criteria for patients:

* Schizophrenic patients as defined in Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV)
* Stabilized a therapeutic point of view for at least one month.
* Consent form signed
* Affiliated to a Security Health Program

Inclusion Criteria for volunteers:

* Consent form signed
* Affiliated to a Security Health Program

Exclusion Criteria for patients and volunteers :

* Not having a history of head trauma, neurological disease or not stabilized serious somatic illness,
* Not to use psychoactive substance, as defined by the DSM IV.
* The Intelligence Quotient must not be less than 70 (Progressive Matrices Standard score (PM38), Raven Progressive Matrix).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2011-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of items recalled TBR and TBF | Day 1
  It is asked to the participants to recall orally, only TBR verbs (task of reminder). The experimenter notes the given verbs.

SECONDARY OUTCOMES:
Number of recognized items | Day 1
  Participants must recognize TBR verbs among several verbs (distractor or TBF verbs) on the screen.The experimenter notes the recognized verbs.
  The recognition of a verb in the TBF list or a distractor is considered like an error.
Reaction time (ms) on the recognition of TBR and TBF | Day 1
  The response times of participants are recorded in ms.

CONTACTS AND LOCATIONS:
Overall Officials: Anne GROSSELIN, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No